CLINICAL TRIAL: NCT03378726
Title: SPOON: Sustained Program for Improving Nutrition - Colombia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inter-American Development Bank (Other)
Collaborators: Fundación Saldarriaga Concha (Other); Instituto Departamental de Salud de Nariño (Unknown); Ministerio de Salud y Protección Social de Colombia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Inter-AmericanDB Colombia
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-02

CONDITIONS: Exclusive Breast Feeding; Child Obesity; Malnutrition, Child
MeSH Terms: conditions — Breast Feeding; Pediatric Obesity; Child Nutrition Disorders | interventions — Micronutrients; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Counseling and Micronutrients (Experimental): Participants will receive standard services provided by the Ministry of Health, including powder micronutrients. Children receive 1 gram of powdered micronutrientes for 60 days between 6 and 12 months of age, and 60 daily packets per year from the time they are 1 year old until 5 years old.
  Interventions: Dietary Supplement: Micronutrients; Behavioral: Standard Counseling
- SPOON Group Counseling with SQ-LNS (Experimental): Participants will receive the supplement SQ-LNS in addition to SPOON group counseling, which is a new form of social communication in which participants will learn relevant lessons in a group format. SQ-LNS consists of a 20g nutrient supplement package that is to be consumed daily between 6 and 24 months of age.
  Interventions: Behavioral: SPOON Group Counseling; Dietary Supplement: SQ-LNS
- Group, Interpersonal Counseling, SQ-LNS (Experimental): Participants will receive the supplement SQ-LNS in addition to SPOON group and interpersonal counseling, which will consist of both participants learning relevant lessons in group format as well as in formats in which participants will work one-on-one with an instructor. SQ-LNS consists of a 20g nutrient supplement package that is to be consumed daily between 6 and 24 months of age.
  Interventions: Behavioral: SPOON Group Counseling; Behavioral: Interpersonal Counseling; Dietary Supplement: SQ-LNS

INTERVENTIONS:
Dietary Supplement: Micronutrients — Micronutrient powder is the current supplement provided by the Colombian Ministry of Health and Social Protection to children between 1 and 5 years of age.
  Arms: Standard Counseling and Micronutrients
Behavioral: SPOON Group Counseling — SPOON group counseling is an innovative behavior change strategy in which participants will learn information related to child health and nutrition in a group format.
  Other Names: Group
  Arms: Group, Interpersonal Counseling, SQ-LNS; SPOON Group Counseling with SQ-LNS
Behavioral: Interpersonal Counseling — SPOON interpersonal counseling is an innovative behavior change strategy in which participants will learn information via one-on-one sessions with the instructor.
  Other Names: SPOON Interpersonal Counseling
  Arms: Group, Interpersonal Counseling, SQ-LNS
Dietary Supplement: SQ-LNS — SQ-LNS is a peanut-based dietary supplement that has been shown to increase children's height and weight in several studies in Africa.
  Other Names: Small Quantity Lipid Nutrient Supplements
  Arms: Group, Interpersonal Counseling, SQ-LNS; SPOON Group Counseling with SQ-LNS
Behavioral: Standard Counseling — Standard counseling refers to the counseling currently provided by health personnel to women and children in the selected intervention area of Colombia
  Arms: Standard Counseling and Micronutrients

SUMMARY:
The primary goal of this study is to prevent undernutrition and obesity in peri-urban areas of Colombia. This study is designed to evaluate the impact of promoting adequate feeding practices and the use of SQ-LNS (Small Quantity Lipid-Based Nutrient Supplements) on the nutritional status of infants and young children. The study will be conducted in peri-urban areas of Pasto, Colombia in conjunction with Fundación Saldarriaga Concha and the Colombian Ministry of Health and Social Protection.

DETAILED DESCRIPTION:
SPOON Colombia is an innovative strategy to prevent undernutrition and obesity in children aged 0-24 months living in high-poverty areas of Colombia. The SPOON program aims to improve infant and young children feeding practices, including exclusive breastfeeding during a child's first six months and home-fortification with peanut-based SQ-LNS (small quantity lipid-based nutrient supplements) for children 6 to 24 months of age.

The SPOON intervention will randomly assign participants at the household level to one of three groups: a control group, Treatment Group 1, and Treatment Group 2. Participants in the control group will receive the standard services provided by their local health clinics in addition to a supply of micronutrient powder. The powder consists of vitamins and minerals that are added to the child's food to increase his or her consumption of micronutrients. Participants in Treatment Group 1 will receive group counseling and the SQ-LNS supplement instead of micronutrient powder. The group counseling program consists of various lessons for the children's caregivers about the importance of breastfeeding and providing high quality food with the SQ-LNS supplement. Those assigned to Treatment Group 2 will receive all the services that those in Treatment Group 1 receive in addition to individualized counseling, where messages about nutrition and breastfeeding will be reinforced through home visits.

Comparing the three treatment arms will identify the marginal impact of the SPOON program. For example, measuring the differences in outcomes between the participants in the control arm and in Treatment Group 1 will identify the impact of the Spoon program package, which includes SQ-LNS and group counseling, compared to current government-provided services. Measuring the differences between Treatment Group 1 and Treatment Group 2 will indicate the marginal impact of individualized counseling, and measuring the difference between the control arm and Treatment Group 2 will determine the combined impact of the SPOON program combined with individualized counseling.

ELIGIBILITY:
Inclusion Criteria:

* Participants must live in the defined intervention areas

Exclusion Criteria:

* Any chronic disease or malformation
* Caretakers of the children plan on moving in the next 24 months

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in Height and Weight from Baseline to 8 months old | Measured when child is 6 months old at baseline and when child is 8 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 8 months old to 10 months old | Measured when child is 8 months old and when child is 10 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 10 months old to 12 months old | Measured when child is 10 months old and when child is 12 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 12 months old to 14 months old | Measured when child is 12 months old and when child is 14 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 14 months old to 16 months old | Measured when child is 14 months old and when child is 16 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 16 months old to 18 months old | Measured when child is 16 months old and when child is 18 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 18 months old to 20 months old | Measured when child is 18 months old and when child is 20 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 20 months old to 22 months old | Measured when child is 20 months old and when child is 22 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject
Change in Height and Weight from 22 months old to 24 months old | Measured when child is 22 months old and when child is 24 months old
  Prevalence of stunting and being overweight, height for age z-score, body mass index z-score will be determined from measuring the height and weight of the subject

SECONDARY OUTCOMES:
Change in Cephalic Circumference from Baseline | Measured when child is 6 months old and when child is 2 years old
  An indicator often used as a proxy for child growth and development
Change in Eating Habits from Baseline | Measured when child is 6 months old and when child is 2 years old
  Include what kinds, quantity, and frequency of food was consumed
Change in Health Status from Baseline | Measured when child is 6 months old and when child is 2 years old
  General health status includes frequency and intensity of diarrhea
Change in Measures of Caregiver Knowledge from Baseline | Measured when child is 6 months old and when child is 2 years old
  Caregiver knowledge in nutrition, hygiene and exclusive breastfeeding will be measured
Change in Prevalence of Anemia from Baseline | Measured when child is 6 months old and when child is 2 years old
  The prevalence of anemia will be measured by reviewing hemoglobin and hematocrit levels
Weight Gain Rate | Measured every 2 months when child is between 6 and 24 months old
  Defined as rate of weight gain of the participating children

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Martinez, Study Director — Inter-American Development Bank

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual data will be shared among participating research institutions and made public 2 years after finalizing the study